CLINICAL TRIAL: NCT02641795
Title: Robotic Assisted Cochlear Implantation Feasibility Study
Acronym: MIRACI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment and extended study duration
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-13-12-011779; PB_2017-0031 (Other: Ethics commision Bern, Switzerland); 2013-MD-0042 (Other: Swissmedic (regulatory authority)); CIV-13-12-011779 (Other: EUDAMED)
Record Dates: First submitted 2015-12-19; First posted 2015-12-29 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Sensory Hearing Loss
Keywords: cochlear implantation; robotics; image guidance
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Minimally invasive robotic cochlear implantation with custom device
  Interventions: Device: Minimally invasive robotic cochlear implantation

INTERVENTIONS:
Device: Minimally invasive robotic cochlear implantation

SUMMARY:
A first in man clinical trial to asses the the use of am image guided robotic system to safely and effectively create a minimally invasive access tunnel to the middle ear cavity to allow access to the round window for cochlear implant electrode insertion.

DETAILED DESCRIPTION:
A first in man feasibility study of an image guided robotic system for performing a key-hole approach to the middle ear cavity.

ELIGIBILITY:
Inclusion Criteria:

* Geographically and physically able to attend scheduled evaluations and follow-up appointments
* Indicated for cochlear implantation
* Age 18 years or older
* Fluent in German or French
* Sufficient facial recess size ( > 2.5 mm between the facial nerve and chorda tympani)

Exclusion Criteria:

* Pregnancy
* Anatomical malformation of the middle or inner ear or unusual facial nerve course
* Lack of compliance with any inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Drilling accuracy | Image data acquired during the procedure
  The lateral distance between the center lines of the planned and drilled tunnel positions at the level of the facial nerve measured from medical image data

SECONDARY OUTCOMES:
Number of successfully completed robotic procedures | The procedure (day 0)
  The number of procedures drilled robotically to the middle ear cavity
The number of successful cochlear implant electrode array insertions | The procedure (day 0)
  Number of electrode arrays implanted through the key-hole approach to the middle ear cavity
Registration accuracy | The procedure (day 0)
  Fiducial matching error of patient to image registration
Time of the robotic procedure and its subparts | The procedure (day 0)
  Total time of the robotic procedure from opening to closing (mean and standard deviation) and of the subprocesses
Adverse events | day 0-30
  Any clinical complications including facial nerve or chorda tympani damage, infection, negative audiological outcomes etc
Blood loss | The procedure (day 0)
  Intraoperative blood loss (ml)
Postoperative pain | day 0-30
  Pain scale and prescribed pain medication
Invasiveness of the intervention | The procedure (day 0)
  Size of incision (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Caversaccio, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital University Hospital Bern, Bern, Switzerland